CLINICAL TRIAL: NCT05907135
Title: Influence of 2-Weeks Beet Pre-Workout Supplement Ingestion on Inflammation Resolution and Metabolic Recovery After Vigorous Exercise
Brief Title: Beet Supplementation, Exercise, Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Standard Process (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-23-297
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Response; Metabolic Disturbance; Immune Suppression
Keywords: Beets; exercise; inflammation; immune function; oxylipins; proteomics
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — Sucrose

STUDY DESIGN:
Intervention Model Description: Randomized treatment, double blinded procedures, crossover
Who Masked: Participant, Investigator
Masking Description: Investigators and study participants will be blind to treatment allocation, with the beet-based supplement and placebo supplement of the same color and taste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beet (Experimental): Powdered beets with green tea extract, Camu Camu, Quinoa sprouts, 3 mushroom blend.
  Interventions: Dietary Supplement: Beet
- Placebo (Placebo Comparator): Similar colored powder with no active ingredients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beet — Beet-based powder with other ingredients
  Arms: Beet
Dietary Supplement: Placebo — Placebo powder.
  Arms: Placebo

SUMMARY:
This study will determine if ingesting a beet-based supplement with nitrates for 2 weeks moderates exercise-induced inflammation.

DETAILED DESCRIPTION:
RESEARCH DESIGN: Subjects will come to the lab for orientation/baseline testing, pre-and post-supplementation blood sample collections (2 weeks supplementation with POSSIBLE Beet Pre-Workout supplement (Standard Process, Kannapolis, NC) or placebo), two 2.25 h cycling sessions, and additional lab visits to provide 1-day 7:00 am recovery blood samples) (thus 7 total lab visits). The total amount of time subjects will be asked to volunteer for this study is about 20 hours at the Human Performance Laboratory (over a 6-week period).

A. Orientation/Baseline Testing (Visit #1) After voluntarily signed IRB-approved consent forms, study participants will be tested for maximal aerobic capacity (VO2max) during a graded, cycling test with continuous metabolic monitoring with the Cosmed CPET metabolic device (Cosmed, Rome, Italy). Body composition will be measured with the seca BIA and Bod Pod body composition analyzer (Life Measurement, Concord, CA). Demographic and training histories will be acquired with questionnaires.

B. Pre-Supplementation Lab Visit #2 and 2-Week Supplementation Protocol: Two weeks prior to the first cycling session, subjects will report to the Human Performance Laboratory at approximately 7:00-8:00 am. A blood sample will be collected in an overnight fasted state to coincide with the same time of the day for the post-supplementation blood draw. A 2-week supply of POSSIBLE Beet Pre-Workout supplement or placebo supplement will be given to the participants. Subjects will mix the supplement powder in one cup of cold water and consume one dose in the early morning and a second dose mid-day.

POSSIBLE Beet Pre-Workout supplement (subjects will consume 2 scoops per day, 28 grams total, with one dose in the early morning, and the second dose mid-day). Note: the placebo will include excipients only, with none of the ingredients listed below.

Ingredients (per 14 g scoop dose) Beets: Beets in combination with fermented beets to provide nitrates (106 mg of nitrates per serving).

Caffeine (100 mg) from Green Tea Extract. Camu Camu to provide vitamin C (22 mg or 25% of the Daily Value). Camu camu is a sour berry native to the Amazon rainforest that has a high vitamin C content.

Quinoa Sprouts: Source of B-vitamins and will provide 20% of the Daily Value for thiamin, riboflavin, niacin, and vitamin B6. Quinoa is a plant with edible seeds that are rich in B vitamins.

Mushroom Blend of three common mushrooms (1.5 g evenly divided from Hericium erinaceus or lion's mane mushroom, Cordyceps sinensis or caterpillar fungus, and Inonotus obliquus or chaga). These three mushrooms may support exercise performance, but more scientific evidence is needed.

C. 2.25 h Cycling Session (Lab Visit #3): During the 3-day period prior to the 2.25-h cycling session, subjects will taper exercise training and ingest a moderate-carbohydrate diet using a food list restricting high fat foods, visible fats, caffeine, and polyphenols (1,2). Study participants will report to the Human Performance Lab in an overnight fasted state and provide a blood sample, ingest the supplement (POSSIBLE Beet Pre-Workout supplement or placebo), and then cycle 2.25 h at high intensity (70% VO2max) while ingesting water alone (3 ml/kg every 15 minutes). Blood samples will be collected at 0 h, 1.5 h, 3.0 h, and 24 h post-exercise.

Testing protocol during the lab sessions with the 2.25-h cycling session:

1. 7:00 am: Provide blood sample, delayed onset of muscle soreness (DOMS) rating (1-10 scale), and profile of mood states ratings (POMS).
2. 7:10 am: Ingest supplement with 1 cup water.
3. 7:30 am: Start the 2.25 h cycling session. Subjects will cycle on trainers at 70% VO2max (~race pace) for 2.25 hours. Oxygen consumption, carbon dioxide production, respiratory exchange ratio, and ventilation will be measured using the Cosmed Quark CPET metabolic cart every 30 minutes. Subjects will consume 3 ml/kg water every 15 min. No other beverage or food containing energy or nutrients will be allowed during the 2.25-h exercise sessions.
4. ~10:00 am to 1:00 pm: Blood samples will be taken via venipuncture immediately after completing the cycling session, and then 1.5-h and 3.0-h post-exercise. Subjects will be allowed to shower and change clothes. The DOMS and POMS questionnaires will be administered each time blood samples are collected. Subjects will ingest no food or beverage other than water (7 ml/kg during the 1.5 h post-exercise period). After the 1.5 h post-exercise blood draw, subjects will ingest a Boost beverage (8 kcal/kg body weight). Another blood sample will be collected 3-h post-exercise. Afterwards, subjects will be allowed to leave the lab with instructions to adhere to the food list requirements, and to keep exercise training moderate.
5. 7:00 am, next morning: 24-h blood sample and DOMS and POMS ratings (Lab visit #4).

D. Washout/Crossover/Repeat Subjects will engage in a 2-week washout period without the supplements, crossover to the opposite treatment arm, and then repeat all procedures (Lab visits #5,6,7).

STATISTICAL ANALYSIS AND POWER CALCULATION The study participant number (N = 20) will provide 84% power to detect a difference with an effect size 0.7 at alpha 0.05 using 2-sided paired t-tests (5). Data will be checked for normality of the residuals using Q-Q plots. All data will be analyzed using the generalized linear model (GLM), and a 2 (condition) x 6 (time) repeated-measures ANOVA, within-participants design (IBM SPSS Statistics for Windows, Version 24.0, IBM Corp, Armonk, NY, USA). Changes over time within conditions will be contrasted between trials using paired t-tests, with the alpha level set at p,0.01. Principle component analysis (PCA) and heatmap analysis of the oxylipin data will be performed with the R programming language (https://www.r-project.org/, version 3.3.1).

ELIGIBILITY:
Inclusion Criteria:

* Male or female cyclists, ages 18-60 years, and capable of cycling 2.25 h in the laboratory at 70% VO2max (close to race pace).
* Non-smoker, and generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis. Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.
* Agree to train normally, maintain weight, and avoid the regular use of large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation (especially NSAIDs) for the duration of the 6-week study and at least a 2-week period prior to the study.
* Agree to limit intake of nitrate-rich vegetables during the study to less than 1 cup per day. These include spinach, lettuce, beets, beetroot juice, celery, and cabbage.
* Agree to taper their exercise routine prior to each of the two lab cycling sessions.
* Agree to avoid the use of mouthwashes, antacids, and chewing gum during the entire 6-week study and the 2-week period prior to the study.

Exclusion Criteria:

* Inability to comply with study requirements.
* Females: body weight below 110 pounds; trying to become pregnant, pregnant or breastfeeding.
* Any other concurrent condition which, in the opinion of the principal investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).
* An unwillingness to avoid mouthwashes, antacids, and chewing gum 2 weeks before and during the 6-week study.
* An unwillingness to limit intake of nitrate-rich vegetables 2 weeks before and during the 6-week study.
* Current history of uncontrolled hypertension and/or the use of vasodilatory medications.
* Sensitivity to caffeine intake from green tea extract (200 mg per day).
* History of allergic reactions to any of the ingredients in the study supplement: beet powder, camu camu, green tea extract, mushroom blend (caterpillar fungus, lion's mane, chaga), quinoa sprouts, monk fruit, pineapple, cranberry seed powder, strawberry fruit powder).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Plasma lipid mediators | Change from pre-study to post-2 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exercise
  Plasma concentrations of arachidonic acid oxidized derivatives from LC-MS/MS analysis

SECONDARY OUTCOMES:
Plasma proteins | Change from pre-study to post-2 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exercise
  Plasma concentrations of immune- and inflammation-related proteins from proteomics profiling using LC-MS/MS.
Plasma nitrate and nitrite concentrations | Change from pre-study to post-2 weeks supplementation, and immediately post-exercise, and 1.5 hours-, and 24 hours-post-exercise
  Plasma concentrations of nitrate and nitrite using ELISA kits

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share data upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2023, indefinitely
Access Criteria: Upon reasonable request.